CLINICAL TRIAL: NCT00004252
Title: A Randomized, Open-Label, Multicenter Phase III Study of 5-FU/Leucovorin With or Without Concomitant SU5416 in Patients With Metastatic Colorectal Cancer
Brief Title: Leucovorin and Fluorouracil With or Without SU5416 in Treating Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: SUGEN-SU5416.031; CDR0000067499; UCLA-9909008
Record Dates: First submitted 2000-01-28; First posted 2004-04-19 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-09

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Fluorouracil; Leucovorin; Semaxinib

INTERVENTIONS:
Drug: fluorouracil
Drug: leucovorin calcium
Drug: semaxanib

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. SU5416 may stop the growth of colorectal cancer by stopping blood flow to the tumor. It is not yet known whether chemotherapy is more effective with or without SU5416 in treating metastatic colorectal cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of leucovorin and fluorouracil with or without SU5416 in treating patients who have metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the median survival in patients with metastatic colorectal cancer treated with fluorouracil and leucovorin calcium with or without SU5416. II. Compare the time to progression, duration of response, and objective response in these patients on these two regimens. III. Compare the percentage 6 month, 9 month, and one year survival of these patients on these two regimens. IV. Compare the time to treatment failure in these patients on these two regimens. V. Determine the health related quality of life of these patients on these two regimens. VI. Compare the palliative and biologic effects of SU5416 in these patients. VII. Determine the safety and tolerability of fluorouracil and leucovorin calcium plus SU5416 in these patients.

OUTLINE: This is a randomized, open label, multicenter study. Patients are stratified according to performance status (ECOG 0 vs 1), site of primary disease (colon vs rectum), measurable or evaluable disease, and prior fluorouracil adjuvant chemotherapy (none vs at least 1 dose). Patients are randomized to one of two treatment arms: Arm I: Patients receive leucovorin calcium IV over 2 hours and fluorouracil IV bolus 1 hour into leucovorin calcium administration weekly for 6 weeks. Arm II: Patients receive leucovorin calcium IV over 2 hours and fluorouracil IV bolus 1 hour into leucovorin calcium administration weekly for 6 weeks, plus SU5416 twice weekly for 8 weeks. Treatment repeats every 8 weeks in the absence of disease progression or unacceptable toxicity. Quality of life is assessed prior to study, at weeks 4 and 8 of each course, and then post study. Patients are followed post study at one month and then every 2 months until death.

PROJECTED ACCRUAL: A total of 710 patients (355 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed, newly diagnosed or recurrent, metastatic colorectal cancer Primary disease was adenocarcinoma of the colon or rectum Bidimensionally measurable or evaluable disease No CNS metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-1 Life expectancy: At least 12 weeks Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 75,000/mm3 Hemoglobin at least 8 g/dL Hepatic: Bilirubin no greater than 2.2 mg/dL AST no greater than 5 times upper limit of normal Renal: Creatinine no greater than 2.0 mg/dL Creatinine clearance at least 50 mL/min Other: Not pregnant Negative pregnancy test Fertile patients must use effective contraception No known allergy to Cremophor or Cremophor based drug products No uncontrolled colon or small bowel disorders No other malignancy within the past 5 years, except: Basal cell skin cancer Carcinoma in situ of the cervix No other acute or chronic medical or psychiatric condition, or laboratory abnormality that would preclude compliance

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior immunotherapy, vaccine therapy, cytokine therapy, or biologic therapy for metastatic disease No prior angiogenesis inhibition therapy (e.g., metalloproteinase inhibitors, thalidomide, anti-VEGF/Flk-1 monoclonal antibody therapy or other experimental drugs acting directly on the VEGF/Flk-1 signaling pathway) Prior antibody therapy, immunotherapy, gene therapy, vaccine therapy, cytokine therapy, or radioimmunotherapy allowed in adjuvant setting only Concurrent epoetin alfa, filgrastim (G-CSF), or sargramostim (GM-CSF) allowed for anemia, neutropenia, or thrombocytopenia No concurrent immunotherapy Chemotherapy: No prior systemic chemotherapy for metastatic disease No prior intra-arterial cytotoxic chemotherapy No more than one prior course of fluorouracil based adjuvant therapy (e.g., intravenous fluorouracil or capecitabine) with the last dose administered at least 6 months ago No prior SU5416 No other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: At least 2 weeks since prior radiotherapy Concurrent localized palliative radiotherapy allowed unless indicative of disease progression Surgery: At least 4 weeks since prior major surgery (not including surgical placement of a venous access device) Prior surgical resection of hepatic metastases allowed Other: No prior investigational therapy for metastatic disease No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-11; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison L. Hannah, MBBS, Study Chair — SUGEN
Locations (26):
- United States (26):
  - Alabama Oncology, LLC, Montgomery, Alabama
  - Office of Richard Shapiro, Benjamin Stafford, and Sharon J. Yee, Arcadia, California
  - Scripps Clinic, La Jolla, California
  - Tower Hematology Oncology Medical Group, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - St. Francis Hospital, San Francisco, California
  - Comprehensive Cancer Care Specialists of Boca Raton, Boca Raton, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Queen's Medical Center, Honolulu, Hawaii
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Cancer Center of Boston, Boston, Massachusetts
  - Michigan State University, East Lansing, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - APN-IMPATH Research Corporation, Fort Lee, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - New York Medical College, Valhalla, New York
  - Presbyterian Healthcare, Charlotte, North Carolina
  - Raleigh Hematology/Oncology Associates - Wake Practice, Raleigh, North Carolina
  - Hematology/Oncology Associates of NE Pennsylvania, P.C., Scranton, Pennsylvania
  - Associates in Oncology & Hematology, Chattanooga, Tennessee
  - Dial Research Associates, Inc., Nashville, Tennessee
  - Presbyterian Hospital of Dallas, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin